CLINICAL TRIAL: NCT00006428
Title: Management of Chronic Pain in Rehabilitation Project I - Management of Chronic Pain in Persons With Spinal Cord Injury
Brief Title: Chronic Pain in Spinal Cord Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NICHD-0120; P01HD033988 (NIH)
Record Dates: First submitted 2000-11-01; First posted 2000-11-02 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2003-03

CONDITIONS: Spinal Cord Injuries; Pain
Keywords: Spinal Cord injury (SCI); Chronic Pain; Amitriptyline
MeSH Terms: conditions — Spinal Cord Injuries; Pain; Chronic Pain | interventions — Amitriptyline

INTERVENTIONS:
Drug: Amitriptyline

SUMMARY:
This trial tests the effectiveness of the drug amitriptyline vs placebo to relieve chronic pain in adults that have had a spinal cord injury.

DETAILED DESCRIPTION:
This double masked placebo-controlled trial will randomize patients (n=100) with a greater than 6 month history spinal cord injury and a greater than 3 month history of associated pain to a daily dose of amitriptyline or placebo for 6 weeks. Patients will be examined before randomization by a study physician or nurse masked to their treatment assignment. They will be assessed by telephone interview before, during treatment, at the end of treatment and 4 months later to assess pain, pain interference with activities, physical and mental health, and number of health care visits for pain.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury six months ago or longer
* Pain for 3 months or longer

Exclusion Criteria:

* History of cardiovascular disease, seizures, or glaucoma
* Currently taking antidepressant medications
* Currently hyperthyroid or taking thyroid medicine
* Currently pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 1996-08; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Cardenas, M.D., Principal Investigator — University of Washington, Department of Rehabilitation
Locations (1):
- University of Washington, Department of Rehabilitation Medicine, Seattle, Washington, United States

REFERENCES:
- [Background] Leijon G, Boivie J. Central post-stroke pain--a controlled trial of amitriptyline and carbamazepine. Pain. 1989 Jan;36(1):27-36. doi: 10.1016/0304-3959(89)90108-5. PMID 2465530
- [Background] Max MB, Culnane M, Schafer SC, Gracely RH, Walther DJ, Smoller B, Dubner R. Amitriptyline relieves diabetic neuropathy pain in patients with normal or depressed mood. Neurology. 1987 Apr;37(4):589-96. doi: 10.1212/wnl.37.4.589. PMID 2436092
- [Background] Sandford PR, Lindblom LB, Haddox JD. Amitriptyline and carbamazepine in the treatment of dysesthetic pain in spinal cord injury. Arch Phys Med Rehabil. 1992 Mar;73(3):300-1. PMID 1543437
- [Background] Cardenas DD, Warms CA, Turner JA, Marshall H, Brooke MM, Loeser JD. Efficacy of amitriptyline for relief of pain in spinal cord injury: results of a randomized controlled trial. Pain. 2002 Apr;96(3):365-373. doi: 10.1016/S0304-3959(01)00483-3. PMID 11973011
- See also: University of Washington, Department of Rehabilitation Medicine, Pain Management Study website — http://depts.washington.edu/rehab/research/chronic.html
- See also: For more information about the National Institute of Child Health and Human Development. — http://www.nichd.nih.gov/